CLINICAL TRIAL: NCT05787496
Title: A Phase 1, Open-Label, Safety, Tolerability, And Efficacy Study of NC525 in Subjects With Advanced Myeloid Neoplasms
Brief Title: A Safety, Tolerability and Efficacy Study of NC525 in Subjects With Advanced Myeloid Neoplasms
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: As a result of program reprioritization and due to the limited clinical activity observed in the Phase 1 trial, the study has been discontinued.
Sponsor: NextCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NC525-01
Record Dates: First submitted 2023-02-08; First posted 2023-03-28 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia; Relapsed or Refractory Chronic Myelomonocytic Leukemia; Relapsed or Refractory Myelodysplastic Syndrome
Keywords: Advanced Leukemia; Leukemia; NC525; PK; AML; MDS; CMML
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 2mg/kg NC525 (Experimental): Subjects received NC525 IV at 2mg/kg bi-weekly (Q2W) for Cycles 1-6, followed by every 4 weeks (Q4W) thereafter.
  Interventions: Drug: NC525
- 2.5mg/kg NC525 (Experimental): Subjects received NC525 IV at 2.5mg/kg weekly (QW) until overall response (e.g., CR, CRh, or CRi) is achieved, at which time they may switch to Q2W dosing. Subjects in Cohort 2 initially received 3mg/kg weekly but dose was reduced to 2.5mg/kg weekly at FDA request due to change in dosing frequency from Q2W to QW.
  Interventions: Drug: NC525
- 4.5mg/kg NC525 (Experimental): Subjects received NC525 IV at 4.5mg/kg weekly (QW) until overall response (e.g., CR, CRh, or CRi) is achieved, at which time they may switch to Q2W dosing.
  Interventions: Drug: NC525
- 9mg/kg NC525 (Experimental): Subjects received NC525 IV at 9mg/kg weekly (QW) until overall response (e.g., CR, CRh, or CRi) is achieved, at which time they may switch to Q2W dosing.
  Interventions: Drug: NC525
- 13.5mg/kg NC525 (Experimental): Subjects received NC525 IV at 13.5mg/kg weekly (QW) until overall response (e.g., CR, CRh, or CRi) is achieved, at which time they may switch to Q2W dosing.
  Interventions: Drug: NC525
- 18mg/kg NC525 (Experimental): Subjects received NC525 IV at 18mg/kg weekly (QW) until overall response (e.g., CR, CRh, or CRi) is achieved, at which time they may switch to Q2W dosing.
  Interventions: Drug: NC525

INTERVENTIONS:
Drug: NC525 — Monoclonal antibody specific for LAIR-1

SUMMARY:
This is an open-label, non-randomized, Phase 1 study to determine the safety and tolerability of NC525. This study will also assess the clinical benefit in subjects with advanced myeloid neoplasms.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is willing to provide written informed consent for the trial.
2. Be ≥ 18 years of age on the day of signing informed consent.
3. Subject has one of the following Myeloid Neoplasms determined by pathology review at the treating institution:

   1. Relapsed or Refractory AML, Note: Active, relapsed, or refractory AML is defined as any one of the following:

      * Primary induction failure, or (PIF) after 2 or more cycles of therapy,
      * First early relapse after a remission duration of fewer than 6 months,
      * Relapse refractory to salvage combination chemotherapy second or subsequent relapse, or
      * Relapsed or refractory AML with at least 5% blasts by bone marrow biopsy or aspirate, or at least 1% blasts in peripheral blood.
   2. Relapsed or Refractory Myelodysplastic syndrome (MDS) after prior hypomethylating agents.

      Note: Subject must have sub-type MDS-EB2 with 10-19% blasts by bone marrow biopsy or aspirate.
   3. Relapsed or Refractory Chronic myelomonocytic leukemia (CMML) with progressive disease or lack of response to hypomethylating agents
4. A male subject must agree to use approved contraception (based on institutional guidelines) and refrain from sperm donation or expecting to father a child, from Screening through the treatment period and for at least 90 days after the last dose of study treatment.
5. A female subject is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP);
   2. A WOCBP agrees to follow approved contraceptive guidance (based on institutional guidelines) from Screening through the treatment period and for at least 90 days after the last dose of study treatment.
6. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
7. Life expectancy greater than or equal to 12 weeks as judged by the Investigator.
8. Have adequate organ function as defined in the protocol.

Exclusion Criteria:

1. Has a diagnosis of acute promyelocytic leukemia (M3, APL), accelerated phase or blast crisis of chronic myeloid leukemia.
2. History or presence of clinically relevant CNS pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis.
3. Patients with active Central Nervous System (CNS) involvement (such as leukemic infiltration, blast in the spinal fluid, or subjects with extramedullary disease).
4. A WOCBP who has a positive pregnancy test (within 72 hours) prior to treatment.
5. History or evidence of any other clinically significant disorder, condition or disease (e.g., symptomatic congestive heart failure, unstable angina pectoris, symptomatic myocardial infection, uncontrolled cardiac arrhythmia, pericardial disease or heart failure New York Heart Association Class III or IV), or severe debilitating pulmonary disease, that would potentially increase patients' risk for toxicity and in the opinion of the Investigator, would pose a risk to patient safety or interfere with the study evaluation, procedures or completion.
6. Chronic respiratory disease or any other medical condition that requires continuous oxygen that in the opinion of the Investigator, would adversely affect his/her participation in this study.
7. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of study intervention.
8. Is currently participating in or has participated in a study of the following prior to the first dose of study treatment:

   1. An investigational biologic or an investigational device within 4 weeks or 5 half-lives (whichever is longer);
   2. An investigational oral agent within 2 weeks or 5 half-lives (whichever is shorter).
9. Has not recovered to ≤ Grade 1 from toxic effects of prior therapy (including prior chemotherapy, immunotherapy and radiation therapy) and/or complications from interventions before starting therapy.
10. Has previously had an allogeneic solid organ transplant.
11. Autologous HSCT within 6 weeks before the start of study treatment.
12. Allogeneic HSCT within 6 months before the start of study treatment.
13. Any active acute or chronic graft-versus-host disease (GvHD), grade 2-4, or active chronic GvHD requiring systemic treatment.
14. Any systemic therapy (e.g. calcineurin inhibitors (CNI), steroids, etc.) against GvHD within 4 weeks before the start of study treatment.
15. Any Grade ≥ 2 persistent non-hematological toxicity related to allogeneic transplant, such as those requiring systemic immunosuppressive therapy.
16. Previous CAR-T therapy.
17. Known concurrent malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry after treatment with curative intent.
18. Has severe hypersensitivity (≥ Grade 3), known allergy or reaction to Immunoglobulins or NC525, and/or any of their excipients.
19. Uncontrolled systemic fungal, bacterial, viral, or other infection despite appropriate anti-infection treatment at the time of eligibility confirmation.
20. Has a known history of HIV infection.
21. Has a known active chronic hepatitis B infection or chronic hepatitis C infection with the exception of those with an undetectable viral load within 3 months.
22. Has a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the study or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate, in the opinion of the treating investigator.
23. Has a known psychiatric or substance abuse disorder that would interfere with the subject's ability to cooperate with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Han Myint, MD, Study Director — NextCure, Inc.
Locations (11):
- United States (11):
  - City of Hope, Duarte, California
  - University of Miami, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medicine, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2mg/kg NC525 | 2.5mg/kg NC525 | 4.5mg/kg NC525 | 9mg/kg NC525 | 13.5mg/kg NC525 | 18mg/kg NC525
Started | 3 | 4 | 3 | 11 | 4 | 3
Completed | 1 | 3 | 2 | 5 | 3 | 1
Not Completed | 2 | 1 | 1 | 6 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Study Terminated by sponsor | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 2 | 1 | 1 | 4 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2mg/kg NC525 | 2.5mg/kg NC525 | 4.5mg/kg NC525 | 9mg/kg NC525 | 13.5mg/kg NC525 | 18mg/kg NC525 | Total
Number analyzed (Participants) | 3 | 4 | 3 | 11 | 4 | 3 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (8.96) | 65.8 (19.87) | 66.0 (10.54) | 69.6 (12.86) | 52.8 (17.97) | 56.7 (24.01) | 64.0 (15.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 2 | 4 | 2 | 1 | 13
  Male | 0 | 3 | 1 | 7 | 2 | 2 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2 | 1 | 1 | 6
  Not Hispanic or Latino | 3 | 2 | 3 | 9 | 3 | 2 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 0 | 0 | 2
  White | 2 | 3 | 3 | 9 | 2 | 2 | 21
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 3 | 11 | 4 | 3 | 28

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate the Frequency, Duration, and Severity of Treatment-emergent Adverse Events [Safety and Tolerability].
Description: Toxicity grading per NCI CTCAE v5.0.
Time Frame: Up to 23 months
Population: Safety Analysis Set (SAS): The SAS will include all the subjects who receive any amount of NC525 and will be used for summaries and analyses of safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | 2mg/kg NC525 | 2.5mg/kg NC525 | 4.5mg/kg NC525 | 9mg/kg NC525 | 13.5mg/kg NC525 | 18mg/kg NC525
Number analyzed (Participants) | 3 | 4 | 3 | 11 | 4 | 3
Participants | 3 | 4 | 3 | 11 | 4 | 3

2. Primary Outcome: To Evaluate Dose-limiting Toxicities (DLTs) of NC525.
Description: Toxicity grading per NCI CTCAE v5.0.
Time Frame: Up to 56 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 2mg/kg NC525 | 2.5mg/kg NC525 | 4.5mg/kg NC525 | 9mg/kg NC525 | 13.5mg/kg NC525 | 18mg/kg NC525
Number analyzed (Participants) | 3 | 4 | 3 | 11 | 4 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: To Evaluate the Clinical Benefit of NC525 by Assessing Objective Response (OR).
Description: Disease Assessments will be performed using the European Leukemia Net (ELN) Guidelines for the ELN Outcome Measures.
Time Frame: Until disease progression, up to 23 months
Population: Full Analysis Set (FAS): The FAS includes all subjects enrolled in the study who received at least one full dose of NC525. The FAS will be used for summaries and analyses of all data that are not safety or PK
Measure: Count of Participants; unit: Participants
Arm/Group | 2mg/kg NC525 | 2.5mg/kg NC525 | 4.5mg/kg NC525 | 9mg/kg NC525 | 13.5mg/kg NC525 | 18mg/kg NC525
Number analyzed (Participants) | 3 | 4 | 3 | 11 | 4 | 3
Participants | 0 | 0 | 0 | 1 | 0 | 0

4. Secondary Outcome: To Evaluate the Clinical Benefit of NC525 by Assessing Event-free Survival (EFS).
Description: Disease Assessments will be performed using the European Leukemia Net (ELN) Guidelines for the ELN Outcome Measures.
Time Frame: Until disease progression, up to 23 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 2mg/kg NC525 | 2.5mg/kg NC525 | 4.5mg/kg NC525 | 9mg/kg NC525 | 13.5mg/kg NC525 | 18mg/kg NC525
Number analyzed (Participants) | 3 | 4 | 3 | 11 | 4 | 3
months | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.

5. Secondary Outcome: To Evaluate the Clinical Benefit of NC525 by Assessing Overall Survival (OS).
Description: Disease Assessments will be performed using the European Leukemia Net (ELN) Guidelines for the ELN Outcome Measures.
Time Frame: Time until death, up to 23 months
Population: Full Analysis Set (FAS): The FAS includes all subjects enrolled in the study who received at least one full dose of NC525. The FAS will be used for summaries and analyses of all data that are not safety or PK. The analysis population includes all participants who received at least one dose of NC525 in each dose cohort. All participants were included in the analysis regardless of whether they experienced the event (death). Overall survival was analyzed using the Kaplan-Meier method.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 2mg/kg NC525 | 2.5mg/kg NC525 | 4.5mg/kg NC525 | 9mg/kg NC525 | 13.5mg/kg NC525 | 18mg/kg NC525
Number analyzed (Participants) | 3 | 4 | 3 | 9 | 2 | 2
months | 3.8 [3.6 to NA] — The upper bound of the 95% confidence interval for the median overall survival could not be estimated due to the very small sample size and limited number of participants in this cohort. Although all participants experienced the event, the Kaplan-Meier variance estimate was insufficient to calculate an upper confidence limit. | 6 [3.1 to NA] — The upper bound of the 95% confidence interval for the median overall survival could not be estimated due to the very small sample size and limited number of participants in this cohort. Although all participants experienced the event, the Kaplan-Meier variance estimate was insufficient to calculate an upper confidence limit. | 6.5 [2.5 to NA] — The upper bound of the 95% confidence interval for the median overall survival could not be estimated due to the very small sample size and limited number of participants in this cohort. Although all participants experienced the event, the Kaplan-Meier variance estimate was insufficient to calculate an upper confidence limit. | 4.1 [1.1 to 7.7] | NA [1.5 to NA] — The median overall survival and corresponding upper confidence interval could not be estimated due to the very small sample size and insufficient information to support Kaplan-Meier estimation. | 3.1 [2.6 to NA] — The upper bound of the 95% confidence interval for the median overall survival could not be estimated due to the very small sample size and limited number of participants in this cohort. Although all participants experienced the event, the Kaplan-Meier variance estimate was insufficient to calculate an upper confidence limit.

6. Secondary Outcome: Assessment of Time to Achieve Response, Defined as CR, CRi, or CRh
Description: Disease Assessments will be performed using the European Leukemia Net (ELN) Guidelines for the ELN Outcome Measures.
Time Frame: Cycle 1 Day 1 to day remission is achieved, up to 23 months (each cycle is 28 days)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 2mg/kg NC525 | 2.5mg/kg NC525 | 4.5mg/kg NC525 | 9mg/kg NC525 | 13.5mg/kg NC525 | 18mg/kg NC525
Number analyzed (Participants) | 3 | 4 | 3 | 11 | 4 | 3
months | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [1.8 to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events.

7. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of NC525
Description: To evaluate the maximum observed serum concentration (Cmax) of NC525. The values reported are Cmax at Cycle 2 Day 1.
Time Frame: During Cycles 1, 2, 3, 5, 7, and 11 (each cycle is 28 days)
Population: The PK analysis set (PAS) will include all the subjects whose blood samples are collected for PK analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | 2mg/kg NC525 | 2.5mg/kg NC525 | 4.5mg/kg NC525 | 9mg/kg NC525 | 13.5mg/kg NC525 | 18mg/kg NC525
Number analyzed (Participants) | 3 | 4 | 3 | 9 | 4 | 3
μg/mL | 26.1 (10.6) | 58.8 (36.5) | 106 (16.3) | 268 (107) | 445 (178) | 585 (176)

8. Secondary Outcome: Terminal Half-life (t1/2) of NC525
Description: To evaluate the Terminal Half-life (t1/2) of NC525.
Time Frame: During Cycles 1, 2, 3, 5, 7, and 11 (each cycle is 28 days), Cycle 1 reported
Population: The PK analysis set includes participants who received NC525 and had sufficient concentration-time data to estimate terminal half-life (t1/2) using noncompartmental analysis. Estimation required an identifiable terminal elimination phase with ≥3 quantifiable post-dose samples. Descriptive statistics were calculated when ≥3 participants had an estimable t1/2. When only 1 participant had an estimable value, the mean is reported and the standard deviation is not calculable.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 2mg/kg NC525 | 2.5mg/kg NC525 | 4.5mg/kg NC525 | 9mg/kg NC525 | 13.5mg/kg NC525 | 18mg/kg NC525
Number analyzed (Participants) | 0 | 3 | 0 | 1 | 1 | 0
h |  | 49.8 (19.6) |  | 55.3 (NA) — Standard deviation is not calculable because only one participant had an estimable terminal half-life (t1/2) value in this Arm/Group. | 64.2 (NA) — Standard deviation is not calculable because only one participant had an estimable terminal half-life (t1/2) value in this Arm/Group. |

9. Secondary Outcome: Area Under the Serum Concentration Versus Time Curve (AUC) of NC525
Description: To evaluate area under the serum concentration versus time curve (AUC) of NC525
Time Frame: During Cycles 1, 2, 3, 5, 7, and 11 (each cycle is 28 days), Cycle 1 reported
Population: The PK analysis set includes participants who received NC525 and had sufficient concentration-time data to estimate AUC using noncompartmental analysis for Cycle 1 Day 1. Participants without adequate quantifiable PK samples were excluded for this parameter. Descriptive statistics were calculated when multiple participants had estimable AUC values. When only one participant had an estimable value, the mean is reported and the standard deviation is not calculable.
Measure: Mean (Standard Deviation); unit: h*μg/mL
Arm/Group | 2mg/kg NC525 | 2.5mg/kg NC525 | 4.5mg/kg NC525 | 9mg/kg NC525 | 13.5mg/kg NC525 | 18mg/kg NC525
Number analyzed (Participants) | 1 | 4 | 3 | 9 | 4 | 3
h*μg/mL | 5540 (NA) — Standard deviation is not calculable because only one participant had an estimable AUC value in this Arm/Group. | 2180 (755) | 5430 (963) | 13000 (4480) | 23900 (8360) | 33700 (19600)

ADVERSE EVENTS:
Time Frame: From first dose of NC525 through 30 days after the last dose (up to approximately 23 months). For SAEs and ECIs from first dose of NC525 through 90 days following cessation of study treatment, or 30 days following cessation of study treatment if the subject initiates new post-treatment cancer therapy, whichever is earlier (up to approximately 23 months).
Arm/Group | 2mg/kg NC525 | 2.5mg/kg NC525 | 4.5mg/kg NC525 | 9mg/kg NC525 | 13.5mg/kg NC525 | 18mg/kg NC525
All-Cause Mortality (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 9/11 | 2/4 | 2/3
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/4 | 2/3 | 9/11 | 4/4 | 3/3
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 11/11 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2mg/kg NC525 (N=3) | 2.5mg/kg NC525 (N=4) | 4.5mg/kg NC525 (N=3) | 9mg/kg NC525 (N=11) | 13.5mg/kg NC525 (N=4) | 18mg/kg NC525 (N=3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 5 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 3 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis fungal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2mg/kg NC525 (N=3) | 2.5mg/kg NC525 (N=4) | 4.5mg/kg NC525 (N=3) | 9mg/kg NC525 (N=11) | 13.5mg/kg NC525 (N=4) | 18mg/kg NC525 (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 6 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 5 | 1 | 1
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 2 | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 2 | 1 | 1
Chills (General disorders) | 1 | 1 | 1 | 2 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 3 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nodule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 3 | 2 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 2 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 1
Cellulitis orbital (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3 | 1 | 2 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Vascular access site haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Vascular access site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Vascular access site swelling (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 2 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Blood lactic acid increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood uric acid decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 3 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 6 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 5 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 4 | 2 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Limb mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 1 | 1
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 1
Differentiation syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 3 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 1 | 3 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 2 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 6 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 3 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 0 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 3 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 1 | 3 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot publish study results before the first multi-center publication. If a multi-center publication is not submitted within 12 months after the end of the study at all sites, or if Sponsor confirms there will be no multi-center publication, the PI may publish study results. However, PI will allow Sponsor at least 30 days to review any publication of study results and Sponsor may request an additional 60 days to review the publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT05787496/Prot_SAP_000.pdf